CLINICAL TRIAL: NCT02289469
Title: PictureRx: Improving Medication Safety in Health Disparity Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PictureRx, LLC (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R44MD004048-04 (NIH)
Record Dates: First submitted 2014-11-09; First posted 2014-11-13 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Medication Reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PictureRx (Experimental): PictureRx medication history platform
  Interventions: Other: PictureRx medication history platform
- Usual care (No Intervention): Usual medication history process

INTERVENTIONS:
Other: PictureRx medication history platform — Tablet PC-based tool to take more complete and accurate medication history
  Arms: PictureRx

SUMMARY:
Medication safety is an important concern in hospital Emergency Departments (EDs), which provide approximately 136 million patient visits annually in the US. An accurate list of the patient's medications is often needed to inform medical decision-making. Moreover, health care facilities are required to provide patients with an accurate, reconciled list of their medications upon completion of the visit. However, for 37-87% of patients in the ED, errors are present in the documented medication list, and patients often leave without an updated list of their medications or a good understanding of their self-care instructions. This increases the risk of harmful adverse drug events. Health disparity populations, who are more likely to seek care in EDs and who more often have difficulty providing a complete medication history, are disproportionately affected.

Health information technology has the potential to improve medication safety in this setting. PictureRx is an internet-based platform designed to improve medication management in vulnerable populations. It allows users to generate illustrated medication lists in an easily-understood, patient-centered format, in either English or Spanish. The investigators have developed a process for importing prescription fill data from the Surescripts Medication History service, which covers 96% of US pharmacies, into the PictureRx platform. The investigators are developing a mobile tablet PC-based medication history platform that receives and processes the Surescripts data, as well as prompts verification and additional information about the medication regimen.

This trial will assess the effect of the PictureRx medication history platform on the accuracy and efficiency of the medication reconciliation process, as well as patient understanding and satisfaction, in hospital Emergency Departments.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed one or more prescription medications

Exclusion Criteria:

* Too ill to complete informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dane Boyington, Ph.D., Principal Investigator — PictureRx, LLC
Locations (1):
- University of Cincinnatti, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 250 patients were enrolled into the intervention group. However, only 244 patients could be matched to suitable controls, and 6 were therefore excluded from the analysis of results. Thus the number of patients recruited was 494 (250 intervention + 244 control), but results are presented for 488 (244 intervention + 244 control).
Groups:
- PictureRx: Participants in the intervention group interacted with the PictureRx medication history platform on a tablet computer to provide information about their medications and verify their list of prescribed medications
- Usual Care: Patients in the usual care group were matched on a 1:1 basis with intervention patients, on the basis of having received care in the same area of the Emergency Department by the same nurse. Their medication information was collected in the usual fashion by interview.
Period: Overall Study
Arm/Group | PictureRx | Usual Care
Started | 250 | 244
Completed | 244 | 244
Not Completed | 6 | 0
Not completed — Unable to match a control | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PictureRx | Usual Care | Total
Number analyzed (Participants) | 244 | 244 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13) | 41 (16) | 41 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 113 | 249
  Male | 108 | 131 | 239
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 144 | 151 | 295
  White or Caucasian | 94 | 71 | 165
  Hispanic | 1 | 13 | 14
  Asian | 0 | 1 | 1
  American Indian or Alaskan Native | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 244 | 244 | 488
ESI acuity level [Count of Participants; unit: Participants] — The Emergency Severity Index (ESI) is a widely-used triage tool, which Emergency Department nurses use to rate patient acuity and resource needs (range 1-5). Briefly, level 1 patients require immediate life-saving intervention. Level 2 are high-risk, have altered mental status, are in severe pain/distress, or may have certain vital sign abnormalities. Level 3 require many resources. Level 4 require one resource. Level 5 require no additional resources. (See www.esitriage.org for more information.)
  Participants
    2 | 32 | 32 | 64
    3 | 102 | 102 | 204
    4 | 96 | 97 | 193
    5 | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes/Updates in Medication List
Description: Participants for whom nurses made updates or corrections to the medication history in electronic health record
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | PictureRx | Usual Care
Number analyzed (Participants) | 244 | 244
Participants | 101 | 43
Statistical Analysis 1: Comparison: PictureRx vs Usual Care; A chi-square test was used to test for differences in proportions between intervention and control groups; Test type: Superiority; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 23.8, 95% CI 2-sided [16.0 to 31.6]

2. Secondary Outcome: Patient Understanding
Description: Assessment of patient understanding of their medication regimen using 4 questions:
  1. I understand what medicines I am supposed to take.
  2. I understand how much medicine I am supposed to take at a time.
  3. I understand what time of day to take each of my medicines.
  4. I understand what each of my medicines is for. Participants had the following response options: Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree Due to formatting restrictions on this site and the results being nearly identical for each question, only answers to question 1 are reported below.
Time Frame: 1 week
Population: A convenience sample of 50 intervention patients was contacted by phone approximately 1 week after Emergency Department discharge to rate their understanding of their medication regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | PictureRx | Usual Care
Number analyzed (Participants) | 50 | 0
Participants
  Strongly Disagree | 0 |
  Disagree | 0 |
  Neutral | 1 |
  Agree | 3 |
  Strongly Agree | 46 |
Statistical Analysis 1: Comparison: PictureRx; Descriptive statistics (counts, frequencies) were used to summarize responses; Test type: Other; p < 0.01, Other

ADVERSE EVENTS:
Arm/Group | PictureRx | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/244
Other Adverse Events (participants affected / at risk) | 0/244 | 0/244

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes